CLINICAL TRIAL: NCT01443091
Title: Oropharyngeal Colostrum for Immune Stimulation in Very Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Children's Miracle Network (Other)
Responsible Party: Principal Investigator, Kristen M. Glass, Assistant Professor of Pediatrics, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CMNPSU-35083
Record Dates: First submitted 2011-09-26; First posted 2011-09-29 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2015-04

CONDITIONS: Very Low Birth Weight Infants
Keywords: very low birth weight infants; VLBW infants; colostrum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colostrum (Experimental)
  Interventions: Other: application of mother's own colostrum
- Sterile water (Placebo Comparator)
  Interventions: Other: application of sterile water

INTERVENTIONS:
Other: application of mother's own colostrum — application of 0.2mL of mother's own colostrum to the infant's oropharyngeal mucosa every 3 hours for 5 days (day of life 2 until day of life 7)
  Arms: Colostrum
Other: application of sterile water — application of 0.2mL sterile water to the infant's oropharyngeal mucosa every 3 hours for 5 days (from day of life 2 until day of life 7)
  Arms: Sterile water

SUMMARY:
Colostrum, mothers' early breastmilk, contains multiple factors that provide immune protection to very low birth weight (VLBW) infants, a population at high risk for hospital-acquired infections. However, critical illness during the first few days of life often prevents the initiation of enteral feeds, placing these infants at even higher risk for morbidities including feeding intolerance and infection. Oropharyngeal administration has been proposed as an alternative route of delivery for colostrum and the immune benefits it provides. Research from animal and adult human models supports oropharyngeal administration as a potentially safe and effective mode of delivery for immune therapies. Immune components of colostrum, such as secretory IgA, may have both direct and indirect effects on the immune system. The purpose of this proposed randomized, placebo-controlled pilot study is to determine the effect of oropharyngeally administered colostrum (OAC) on immune stimulation in VLBW infants, as measured by secretory IgA (sIgA) levels. In addition to measuring sIgA response to OAC the investigators will also collect clinical data to determine if OAC has effects on tolerance of enteral feedings and rates of infection. The investigators hypothesize OAC will have a moderate effect on salivary secretory IgA concentration in VLBW infants. If proven efficacious, utilization of OAC in VLBW infants could have far reaching consequences for these highly fragile babies including lower rates of infection, improved tolerance of enteral feedings, and shorter NICU stays.

ELIGIBILITY:
Inclusion Criteria:

* infants with a birth weight less than 1500 grams (or 3.3 lbs) born at Penn State Hershey Medical Center and admitted to the PSUCH NICU immediately after birth

Exclusion Criteria:

* Infants with major congenital anomalies or chromosomal syndromes incompatible with life Infants of mothers not willing to provide colostrum for their infant in the first week of life Infants of mothers with known HIV, Hepatitis B or Hepatitis C as these infections may be transmitted through breast milk

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in salivary secretory Ig-A concentration from baseline to 2 weeks of age | 2 weeks of age

SECONDARY OUTCOMES:
time to reach full enteric feeds | first few weeks of age
  day of life when full enteral feeds attained, defined as a volume of 140-150mL/kg/day
episodes of suspected or culture positive sepsis | initial hospital stay 1-3 months
  number of documented septic events either culture proven or those treated with a full course of antibiotics 7-14 days

CONTACTS AND LOCATIONS:
Overall Officials: Kristen M Glass, MD, Principal Investigator — Penn State Milton S. Hershey Medical Center/Penn State College of Medicine
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States